CLINICAL TRIAL: NCT05406167
Title: Prospective Data Registry and Quality of Life Assessment of PatientsUndergoing Radiotherapy With the RefleXion Medical Radiotherapy System (PREMIER Registry)
Brief Title: Prospective Data Registry and Quality of Life Assessment of Patients Undergoing Radiotherapy With the RefleXion Medical Radiotherapy System
Acronym: PREMIER
Status: Recruiting | Type: Observational
Sponsor: RefleXion Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 985-00003
Record Dates: First submitted 2022-05-02; First posted 2022-06-06 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Cancer Central Nervous System; Cancer Thoracic; Cancer, Gastrointestinal; Cancer Gynecologic; Cancer, Genito-Urinary; Cancers Lymphatic; Cancer Head and Neck
Keywords: IMRT; SBRT; Radiation Oncology
MeSH Terms: conditions — Neoplasms; Central Nervous System Neoplasms; Gastrointestinal Neoplasms; Urogenital Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Stereotactic Body Radiotherapy [SBRT]: Patients treated with Reflexion X1 with SBRT as the standard of care
  Interventions: Device: Registry - Observational
- Intensity -Modulated Radiation Therapy [IMRT]: Patients treated with Reflexion X1 with IMRT as the standard of care
  Interventions: Device: Registry - Observational
- Biology-guided Radiotherapy [BgRT]: Patients treated with Reflexion X1 with BgRT as the standard of care
  Interventions: Device: Registry - Observational

INTERVENTIONS:
Device: Registry - Observational — Observation Registry for Medical Device
  Other Names: Reflexion X1

SUMMARY:
The purpose of this prospective cohort study is to assess clinical and quality of life measures as well as to define the severity of adverse effects for the use of the RefleXion system to deliver intensity-modulated radiotherapy (IMRT), stereotactic body radiotherapy (SBRT), or SCINTIX Biology-guided radiotherapy (BgRT) in standard of care (SOC) use in the treatment of local,loco-regionally advanced, and oligometastatic malignancies. In addition, patient costs and charges will be analyzed to quantify the health economic impact of this modality. Workflow and quality of radiotherapy planning including a collection of dosimetric data will also be analyzed.

DETAILED DESCRIPTION:
This multi-center prospective registry is designed to assess the efficacy of IMRT, SBRT, and BgRT delivered via the RMRS. The study will seek to enroll approximately 750 patients initially and then remain open to further patients beyond at the discretion of the study sponsor and participating institutions. The number of IMRT, SBRT, and BgRT patients expected to enroll for the initial period is as follows:

* N = 250 IMRT
* N - 250 SBRT
* N - 250 BgRT

Patients diagnosed with local, locoregionally advanced, or metastatic malignancies will be treated with IMRT, SBRT, or BgRT using the RMRS, with total dose, fractionation, and concurrent systemic therapy delivered according to the direction of the radiation oncology care team. The target population is patients for whom standard radiotherapy is prescribed using IMRT, SBRT, and BgRT. Data will be stratified by common radiotherapy divisions as follows:

* Central Nervous System (Brain, spinal cord, and vertebral column)
* Head and Neck
* Thoracic
* Gastrointestinal
* Gynecologic
* Genitourinary
* Lymphoma
* Melanoma/Sarcoma/Extremity
* Non-Spine Bone and Other An additional sub-stratum within each anatomic division will specify whether the treatment intent is for definitive treatment of the primary tumor (for early-stage or locally advanced disease), a definitive oligo/polymetastatic therapy, or a palliative therapy. Patients will be routinely assessed during their radiation course and thereafter for toxicity burden and HRQOL using the CTCAE v5, EORTC, and EuroQOL surveys. Patients will be assessed for 2 years following their therapy. Other long-term follow-ups will capture data including standard of care (per physician's discretion) laboratory evaluation, quality of life questionnaires, performance status, routine radiographic assessments, physical exams, etc. (see Appendix B. Schedule of Events).

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and be willing to sign an informed consent form (ICF).
* Diagnosis of local, loco-regionally advanced, or metastatic malignancy for whom radiotherapy is indicated
* Radiotherapy to be delivered on the RMRS X1 with IMRT, SBRT, or BgRT technique.
* Absence of concurrent illness that deems radiotherapy a contraindication which will be determined by the treating radiation oncologist.
* Female and male patients of child-bearing potential willing to take appropriate precautions to avoid pregnancy while being treated. Permitted methods in preventing pregnancy should be communicated to the patient and their understanding confirmed by the treating Physician.
* For BgRT patients only: Deemed eligible for BgRT with FDG per BgRT planning session

Exclusion Criteria:

* Pregnant or expecting to conceive during the study.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with study requirements and follow-up visits.
* Inability to maintain immobilization, supine position for planning and treatments.
* For BgRT patients only: Known allergy to FDG

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The purpose of this prospective cohort study is to assess clinical and quality of life measures as well as to define the severity of adverse effects for the use of the RefleXion system to deliver intensity-modulated radiotherapy (IMRT), stereotactic body radiotherapy (SBRT), and Biology-guided radiotherapy (BgRT), in standard of care(SOC)use in the treatment of local, locoregionally advanced, and oligometastaticmalignancies. In addition, patient costs and charges will be analyzed to quantify the health economic impact of this modality. Workflow and quality of radiotherapy planning including collection of dosimetric data will also be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQOL) scores | 30 Days
  Evaluate patient-reported quality of life after IMRT, SBRT, or BgRT treatment delivered by the RefleXion system by assessing EORTC QLQ-C30.
  The EORTC questionnaire has a scoring of 0 to 100 and is disease-specific. 0 is none/minimal symptoms and normal/good functional ability. 100 is increased/severe symptoms and decrease/poor functional ability.
Health Related Quality of Life (HRQOL) scores | 90 Days
  Evaluate patient-reported quality of life after IMRT or SBRT treatment delivered by the RefleXion system by assessing EORTC QLQ-C30.
  The EORTC questionnaire has a scoring of 0 to 100 and is disease-specific. 0 is none/minimal symptoms and normal/good functional ability. 100 is increased/severe symptoms and decrease/poor functional ability.

SECONDARY OUTCOMES:
Long Term Health-Related Quality of Life-EORTC | 6 months, 9 months, 12 months, 18 months, and 24 months
  Long-term Health-Related Quality of Life (HRQOL) scores, including the EORTC QLQ-C30 at 6 months, 9 months, 12 months, 18 months, and 24 months.
  The EORTC questionnaire has a scoring of 0 to 100 and is disease-specific. 0 is none/minimal symptoms and normal/good functional ability. 100 is increased/severe symptoms and decrease/poor functional ability.
Long Term Health Related Quality of Life-EuroQol | 6 months, 9 months, 12 months, 18 months, and 24 months
  The EuroQOL-5D-FL (EQ-5D) will be used in parallel with the Health-Related Quality of Life (HRQOL) surveys to measure quality-adjusted life years.
  The EQ-5D comprises five questions on mobility, self-care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.
Acute toxicities related to Radiotherapy treatment | Up to 90 days
  Proportion of patients with acute treatment toxicity for the anatomic site undergoing treatment
Disease Status [progression-free survival] | Through Study Completion, average of 2 years
  Evaluate progression-free survival after intensity-modulated radiotherapy or stereotactic body radiotherapy for the cancers above. For prostate cancer cohort, biochemical progression-free survival will also be measured.
Disease Status [local recurrence] | Through Study Completion, average of 2 years
  Evaluate local control after intensity-modulated radiotherapy or stereotactic body radiotherapy for the cancers above.
Disease Status [regional recurrence] | Through Study Completion, average of 2 years
  Evaluate regional control after intensity-modulated radiotherapy or stereotactic body radiotherapy for the cancers above.
Disease Status [distant recurrence] | Through Study Completion, average of 2 years
  Evaluate distant control after intensity-modulated radiotherapy or stereotactic body radiotherapy for the cancers above.
Disease Status [overall survival] | Through Study Completion, average of 2 years
  Evaluate overall survival after intensity modulated radiotherapy or stereotactic body radiotherapy for the cancers above.
Intervention and Episodic costs | Up to 6 months
  Analyze resource utilization associated with the RefleXion system for the tumors above including the acute costs of intervention & 6-month episodic costs.
Long-term toxicities related to Radiotherapy | After 90 days through study completion
  Analyze long term treatment toxicity for the anatomic site undergoing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sean Shirvani, MD, Study Director — RefleXion Medical; Karine Feghali, MD, Study Director — RefleXion Medical
Locations (5):
- United States (5):
  - City Of Hope, Duarte, California
  - Stanford Cancer Center, Palo Alto, California
  - Yale University - Cancer Center, New Haven, Connecticut
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No